CLINICAL TRIAL: NCT00912184
Title: Pilot Randomised Controlled Study Comparing The Effect of High Cut-off Point Haemofiltration With Standard Haemofiltration In Patients With Acute Renal Failure
Brief Title: Study Comparing High Cut-off Haemofiltration With Standard Haemofiltration in Acute Renal Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rafidah Atan, PhD student, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: High cut-off trial
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Failure, Acute; Shock
Keywords: Kidney failure, acute; Shock; Toxins, biological; Hemofiltration; High cut off/super high flux membranes
MeSH Terms: conditions — Acute Kidney Injury; Shock

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): CVVH with high cut-off polyamide membrane (P2SH) using standard continuous veno-venous hemofiltration (CVVH) settings
  Interventions: Device: High cut-off (super high flux) polyamide membrane
- 2 (Active Comparator): CVVH using standard high flux membrane with standard CVVH settings
  Interventions: Device: Standard polyamide high flux membrane

INTERVENTIONS:
Device: Standard polyamide high flux membrane — Standard haemofiltration; CVVH; blood flow 200 ml/min, ultrafiltrate 25 ml/kg/hr, anticoagulation as clinically indicated, bicarbonate buffered replacement fluid
  Other Names: High flux membrane
  Arms: 2
Device: High cut-off (super high flux) polyamide membrane — CVVH with standard haemofiltration settings; blood flow 200 ml/min, ultrafiltrate 25 ml/kg/hour, anticoagulation as clinically indicated, bicarbonate-buffered replacement fluid
  Other Names: P2SH; Super high flux membrane
  Arms: 1

SUMMARY:
This trial aims to study the effect of combining continuous and a new polyamide membrane with larger pores in the treatment of critically ill patients with acute renal failure and low blood pressure (shock) requiring noradrenaline. The investigators wish to compare the clinical effect of this new therapy to that of haemofiltration with a standard membrane.

DETAILED DESCRIPTION:
During acute renal failure, small and middle molecular-weight toxins accumulate. These molecules are difficult to remove by standard haemofiltration. Accordingly, they accumulate and contribute to morbidity in long-term dialysis patients. Molecules such as cytokines have been shown to play a central pathogenic role in critical illness. In critically ill acute renal failure patients, they accumulate in serum and likely contribute to much morbidity (fever, low blood pressure, myocardial dysfunction, renal failure itself etc.) Therefore, the removal of cytokines appears desirable. Although different approaches have been undertaken, all have had limited success due to complexity, limited efficacy or uncertain clinical response [10-15].

It is possible that in using a different and more porous membrane, the removal of cytokines would be much more efficient and that clinical benefits of blood purification would, therefore, be greater.

A membrane of this kind is now available. It is a modification (moderate increase in pore size) of another standard material called polyamide, which has already been used in millions of people for dialysis and haemofiltration. The increased pore size of these new membranes is directed at a more effective removal of middle molecular-weight toxins such as cytokines.

ELIGIBILITY:
Inclusion Criteria:

* The treating clinician believes that the patient requires haemofiltration for acute renal failure
* The patient is on noradrenaline infusion for haemodynamic support
* The patient was commenced on noradrenaline or haemofiltration within the last 12 hours
* The clinician is uncertain about the balance of benefits and risks likely to be conferred by treatment with different membranes
* The treating clinicians anticipate treating the patient with haemofiltration for at least 72 hours
* Informed consent has been obtained
* The patient fulfils ONE of the following clinical criteria for initiating haemofiltration:
* Oliguria (urine output < 100 ml/6 hr) that has been unresponsive to fluid resuscitation measures.
* Hyperkalemia ([K+] > 6.5 mmol/L)
* Severe acidemia (pH < 7.2)
* Urea > 25 mmol/liter
* Creatinine > 300 mmol/L
* Clinically significant organ oedema in the setting of ARF (e.g., lung)

Exclusion Criteria:

* Patient age is < 18 years
* Death is imminent (< 24 hours)
* There is a strong likelihood that the study treatment would not be continued in accordance with the study protocol
* The patient has been treated with haemofiltration or other dialysis previously during the same hospital admission
* The patient was on maintenance dialysis prior to the current hospitalisation
* Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study
* The patient is pregnant or is breastfeeding
* The patient has previously been enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is noradrenaline free time in the first week after randomization | 24 months

SECONDARY OUTCOMES:
The change in the levels of each of three key cytokines; IL-1, IL-6 and IL-10 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafidah Atan, MBBS, FANZCA, Principal Investigator — Austin Health
Locations (1):
- Austin Hospital, Heidelberg, Victoria, Australia

REFERENCES:
- [Background] Ronco C, Tetta C, Mariano F, Wratten ML, Bonello M, Bordoni V, Cardona X, Inguaggiato P, Pilotto L, d'Intini V, Bellomo R. Interpreting the mechanisms of continuous renal replacement therapy in sepsis: the peak concentration hypothesis. Artif Organs. 2003 Sep;27(9):792-801. doi: 10.1046/j.1525-1594.2003.07289.x. PMID 12940901
- [Background] Marshall JC. Inflammation, coagulopathy, and the pathogenesis of multiple organ dysfunction syndrome. Crit Care Med. 2001 Jul;29(7 Suppl):S99-106. doi: 10.1097/00003246-200107001-00032. PMID 11445742
- [Background] Parrillo JE. Pathogenetic mechanisms of septic shock. N Engl J Med. 1993 May 20;328(20):1471-7. doi: 10.1056/NEJM199305203282008. No abstract available. PMID 8479467
- [Background] Bone RC. Sir Isaac Newton, sepsis, SIRS, and CARS. Crit Care Med. 1996 Jul;24(7):1125-8. doi: 10.1097/00003246-199607000-00010. No abstract available. PMID 8674323
- [Background] Pinsky MR, Vincent JL, Deviere J, Alegre M, Kahn RJ, Dupont E. Serum cytokine levels in human septic shock. Relation to multiple-system organ failure and mortality. Chest. 1993 Feb;103(2):565-75. doi: 10.1378/chest.103.2.565. PMID 8432155
- [Background] Hack CE, Aarden LA, Thijs LG. Role of cytokines in sepsis. Adv Immunol. 1997;66:101-95. doi: 10.1016/s0065-2776(08)60597-0. No abstract available. PMID 9328641
- [Background] Dinarello CA. Proinflammatory cytokines. Chest. 2000 Aug;118(2):503-8. doi: 10.1378/chest.118.2.503. PMID 10936147
- [Background] Glauser MP. The inflammatory cytokines. New developments in the pathophysiology and treatment of septic shock. Drugs. 1996;52 Suppl 2:9-17. doi: 10.2165/00003495-199600522-00004. PMID 8869831
- [Background] Bellomo R, Tipping P, Boyce N. Continuous veno-venous hemofiltration with dialysis removes cytokines from the circulation of septic patients. Crit Care Med. 1993 Apr;21(4):522-6. doi: 10.1097/00003246-199304000-00011. PMID 8472571
- [Background] Bellomo R. Continuous hemofiltration as blood purification in sepsis. New Horiz. 1995 Nov;3(4):732-7. PMID 8574604
- [Background] De Vriese AS, Colardyn FA, Philippe JJ, Vanholder RC, De Sutter JH, Lameire NH. Cytokine removal during continuous hemofiltration in septic patients. J Am Soc Nephrol. 1999 Apr;10(4):846-53. doi: 10.1681/ASN.V104846. PMID 10203370
- [Background] Hoffmann JN, Hartl WH, Deppisch R, Faist E, Jochum M, Inthorn D. Hemofiltration in human sepsis: evidence for elimination of immunomodulatory substances. Kidney Int. 1995 Nov;48(5):1563-70. doi: 10.1038/ki.1995.448. PMID 8544415
- [Background] Gasche Y, Pascual M, Suter PM, Favre H, Chevrolet JC, Schifferli JA. Complement depletion during haemofiltration with polyacrilonitrile membranes. Nephrol Dial Transplant. 1996 Jan;11(1):117-9. PMID 8649617
- [Background] Kellum JA, Johnson JP, Kramer D, Palevsky P, Brady JJ, Pinsky MR. Diffusive vs. convective therapy: effects on mediators of inflammation in patient with severe systemic inflammatory response syndrome. Crit Care Med. 1998 Dec;26(12):1995-2000. doi: 10.1097/00003246-199812000-00027. PMID 9875910
- [Background] Cole L, Bellomo R, Hart G, Journois D, Davenport P, Tipping P, Ronco C. A phase II randomized, controlled trial of continuous hemofiltration in sepsis. Crit Care Med. 2002 Jan;30(1):100-6. doi: 10.1097/00003246-200201000-00016. PMID 11902250
- [Background] Lee WC, Uchino S, Fealy N, Baldwin I, Panagiotopoulos S, Goehl H, Morgera S, Neumayer HH, Bellomo R. Super high flux hemodialysis at high dialysate flows: an ex vivo assessment. Int J Artif Organs. 2004 Jan;27(1):24-8. doi: 10.1177/039139880402700106. PMID 14984180
- [Background] Uchino S, Bellomo R, Morimatsu H, Goldsmith D, Davenport P, Cole L, Baldwin I, Panagiotopoulos S, Tipping P, Morgera S, Neumayer HH, Goehl H. Cytokine dialysis: an ex vivo study. ASAIO J. 2002 Nov-Dec;48(6):650-3. doi: 10.1097/00002480-200211000-00013. PMID 12455777
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Atan R, Peck L, Prowle J, Licari E, Eastwood GM, Storr M, Goehl H, Bellomo R. A Double-Blind Randomized Controlled Trial of High Cutoff Versus Standard Hemofiltration in Critically Ill Patients With Acute Kidney Injury. Crit Care Med. 2018 Oct;46(10):e988-e994. doi: 10.1097/CCM.0000000000003350. PMID 30074491